CLINICAL TRIAL: NCT03268889
Title: Chidamide With Cyclophosphamide, Etoposide, Vincristine and Prednisone for de Novo Peripheral T Cell Lymphoma Patients
Brief Title: Chidamide With CHOP Regimen for de Novo PTCL Patients (CHOP: Cyclophosphamide, Etoposide, Vincristine and Prednisone; PTCL: Peripheral T Cell Lymphoma)
Acronym: CHOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jinzm 001
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Chidamide, CHOP regimen
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; VAP-cyclo protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): In this arm, patients would be given the regimen composed of Chidamide, Cyclophosphamide, epirubicin, Vincristine and Prednisone.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide is given to the patients in this study along with CHOP regimen, to access the efficacy and safety in this cohort of PTCL patients. The dosage of the above regimen is as follows: Chidamide, 30mg,po,biw; Cyclophosphamide 750mg/m2, ivgtt, d1; Epirubicin 70mg/ m2, ivgtt, d1; Vincristine 3mg/ m2, ivgtt, d1; Prednisone 100mg/ m2, po, d1-5.
  Other Names: CHOP regimen

SUMMARY:
This study evaluates the efficacy and safety of Chidamide plus CHOP regimen for de novo PTCL patients.

DETAILED DESCRIPTION:
After enrollment, patients in this study will be given Chidamide, Cyclophosphamide, Epirubicin, Vincristine and Prednisone, and the efficacy and safety of this regimen are then evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed as peripheral T cell lymphoma (PTCL) according to WHO 2008 classification criteria（NK/T cell lymphoma, ALK positive anaplastic large cell lymphoma and granuloma fungoides excluded）;
2. De novo peripheral T cell lymphoma patients;
3. Age 18-70 years old;
4. ECOG≤2；
5. Female patients not in lactation nor pregnancy, and no intention to concept during the study and 12 months thereafter. Male patients agree not to impregnate his partner during the study and 12 months thereafter;
6. The patient should have evaluable foci (lymphnodes with diameter≥1.0cm, or evaluable skin foci);
7. Willing to sign a written consent.

Exclusion Criteria:

1. T lymphoblast lymphoma;
2. Bone marrow infiltrated with lymphoma cell ≥25%；
3. NT/T cell lymphoma;
4. Granuloma fungoides;
5. Severe impaired liver/ renal function (ALT, Bilirubin or creatinine >3 times the normal maximum);
6. Uncontrolled infection;
7. Organic cardiopathy with clinical manifestation or impaired cardiac function (NYHA ≥ level 2);
8. With other tumors;
9. With other condition that cause the patient unable to sign the written consent;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate | every 3 months until 30 months after the last patient's enrollment
  the rate of patients who achieve complete remission after the treatment

SECONDARY OUTCOMES:
progression free survival | from the day of treatment to the date of first documented progression，up to 30 months after the last patient's enrollment
  from date of inclusion to date of progression, relapse, or death from any cause
duration of remission | from the day of treatment to the date of first documented progression，up to 30 months after the last patient's enrollment
  from date of complete remission to date of progression, relapse, or death from any cause
overall survival | 30 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause
adverse events | from the date of first cycle of treatment to 30 months after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zhengming Jin, MD,PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available at the First Affiliated Hospital after the study is finished
Supporting Information: Study Protocol, CSR
Time Frame: From the time of study finish

REFERENCES:
- [Derived] Zong X, Yang Z, Zhou J, Jin Z, Wu D. Clinical trial: Chidamide plus CHOP improve the survival of newly diagnosed angioimmunoblastic T-cell lymphoma. Front Immunol. 2024 Aug 20;15:1430648. doi: 10.3389/fimmu.2024.1430648. eCollection 2024. PMID 39229263